CLINICAL TRIAL: NCT07005999
Title: The Safety and Efficacy of Interventional Ablation for High-risk Pulmonary Nodules or Early-stage Lung Cancer: A Multicenter, Prospective, Real-World Study
Brief Title: Interventional Ablation for Early-stage Lung Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Collaborators: Hunan Provincial People's Hospital (Other); Beijing Chao Yang Hospital (Other); Fuda Cancer Hospital, Guangzhou (Other); University of South China Affiliated Nanhua Hospital (Unknown); Nanfang Hospital, Southern Medical University (Other); The First Affiliated Hospital of Guangzhou Medical University (Other); Sir Run Run Shaw Hospital (Other); Eastern Theater General Hospital,QinHuai District Medical Area (Unknown); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other); Emergency General Hospital (Other); The First Affiliated Hospital of Anhui Medical University (Other); The Second Hospital of Anhui Medical University (Other); Huaxi Hospital (Other); Shanghai Chest Hospital (Other); Military 301 Hospital (Unknown); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Zhou Chengzhi, doctor, Guangzhou Institute of Respiratory Disease
Other Study IDs: CROC-25-02; ES-2025-064-01 (Other: Guangzhou Institute of Resoiratory Health)
Record Dates: First submitted 2025-05-19; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Lung Cancer (NSCLC); Early Stage Lung Non-Small Cell Carcinoma
Keywords: Intercentional Ablation; Early stage lung cancer; Real-world study
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposure Group(A): Subjects were entered into the exposure group because they chose interventional ablation therapy and agreed to be enrolled in this real-world study.
- Control Group(B): Subjects were entered into the control group because they chose surgical resection treatment and agreed to be enrolled in this real-world study.

SUMMARY:
What is this study about? This clinical trial aims to compare two treatments for high-risk lung nodules or early-stage lung cancer: interventional ablation (a minimally invasive procedure that destroys tumors with heat or cold) and surgical resection (surgery to remove the tumor). The goal is to determine if ablation is as safe and effective as surgery while preserving more lung function.

Why is this important? Lung cancer is a leading cause of cancer deaths worldwide. Early detection improves survival, but surgery can damage lung function.

Ablation (e.g., microwave, cryotherapy) is less invasive than surgery and may offer similar outcomes with faster recovery. However, more evidence is needed to confirm its role in early-stage disease.

DETAILED DESCRIPTION:
What is this study about? This clinical trial aims to compare two treatments for high-risk lung nodules or early-stage lung cancer: interventional ablation (a minimally invasive procedure that destroys tumors with heat or cold) and surgical resection (surgery to remove the tumor). The goal is to determine if ablation is as safe and effective as surgery while preserving more lung function.

Why is this important? Lung cancer is a leading cause of cancer deaths worldwide. Early detection improves survival, but surgery can damage lung function.

Ablation (e.g., microwave, cryotherapy) is less invasive than surgery and may offer similar outcomes with faster recovery. However, more evidence is needed to confirm its role in early-stage disease.

Who can participate? Adults aged 20-79 with high-risk lung nodules or early lung cancer.

Eligibility criteria:

Nodules ≤2 cm on CT scan, no lymph node/distant spread. Good overall health (e.g., normal blood/organ function, no severe heart/lung disease).

No recent cancer treatments (e.g., chemotherapy, radiation). Exclusions: Nodules near major blood vessels/chest wall, pregnancy, or uncontrolled medical conditions.

What does the study involve?

Two treatment groups:

Ablation group: Destroy tumors using heat (microwave) or cold (cryoablation). Surgery group: Remove tumors via standard surgery. Follow-up: Regular check-ups for 5 years, including CT scans, lung function tests, and blood work.

What are the potential risks? Ablation risks: Pain, bleeding, infection, pneumothorax (collapsed lung), or damage to nearby organs.

Surgery risks: Infection, prolonged pain, lung complications (e.g., reduced function), or longer recovery.

Both groups may experience recurrence or side effects like fatigue. What are the benefits? Direct benefits: Access to advanced treatments, close monitoring, and potential lung function preservation with ablation.

Long-term impact: Help future patients by improving treatment options for early lung cancer.

Study Timeline and Locations Duration: 2024-2028 (participants followed for up to 5 years). Locations: 18+ major hospitals across China, including Guangzhou Medical University Affiliated Hospital (lead center), West China Hospital, and Shanghai Chest Hospital.

Key Outcomes Measured Relapse-free survival: Time without cancer returning. Safety: Rates of complications (e.g., bleeding, infection). Lung function: Preserved breathing capacity after treatment. Quality of life: Physical and emotional well-being post-treatment. How will results be used? Findings will guide doctors in choosing the best treatment for early lung cancer, balancing effectiveness with quality of life. Results will be published in medical journals and shared at conferences.

Contact Information

For questions or enrollment:

Lead Researcher: Dr. Zhou Chengzhi, Respiratory Medicine, Guangzhou Medical University Affiliated Hospital.

Local Sites: Contact participating hospitals listed in the study document. Ethical Approval: This study follows strict ethical guidelines to protect participants. All treatments are voluntary, and participants may withdraw at any time.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 20-79 years;
2. Eastern Cooperative Oncology Group Physical Status (ECOG PS) score of 0-2;
3. Enhanced CT of the chest: suspicious malignant signs of lung nodules, such as lobar sign, burr sign, pleural depression sign, bronchial insufflation sign, vacuolar sign, vascular cluster sign, or signs of twisted dilatation of blood vessels within the nodule and cystic cavity type, with no more than 3 lesions bilaterally or unilaterally, and no lymph node metastasis;
4. Thin-section CT of the chest: maximum diameter of the lesion > 5mm ≤ 2cm, solid/tumour ratio CTR ≤ 0.25;
5. Adequate haematological, renal and hepatic functions:

   1. Haematology: absolute neutrophil count (ANC) ≥1.5×109/L, platelet (PLT) ≥100×109/L, haemoglobin (HGB) ≥9 g/dL;
   2. Liver function: serum total bilirubin (TBIL) ≤1.5 times the upper limit of normal (ULN), alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≤2.5 times the ULN, serum albumin (ALB) ≥2.8 g/dL;
   3. Renal function: serum creatinine (Cr) ≤ 1.5 x ULN, or creatinine clearance ≥ 40 mL/min;
6. Subjects and subject sexual partners are required to use a medically approved contraceptive method (e.g., IUD, birth control pills, or condoms, etc.) during the study treatment period and for 6 months after the end of the study treatment period; (7) Subjects must sign a written informed consent form approved by the IRB/IEC in accordance with competent authorities and study site guidelines, and be able to comply with protocol-specified visits, treatment regimens, laboratory investigations, and related procedures.

Haematology Neutrophils (ANC) ≥1.5 x 109/L Platelets (PLT) ≥100×109/L Haemoglobin (Hb) ≥90g/L Liver Function Total bilirubin (TBIL) ≤1.5 x upper limit of normal (ULN) Glutamate aminotransferase (ALT) ≤2.5 × ULN; for patients with liver metastases ≤5 × ULN; Aspartate aminotransferase (AST) ≤2.5 x ULN; for patients with liver metastases ≤5 x ULN; Renal function Creatinine (Cr) ≤1.5×ULN; if >1.5×ULN, creatinine clearance ≥50 mL/min (calculated according to the Cockcroft-Gault formula) Coagulation Activated partial thromboplastin time (APTT) ≤1.5×ULN Prothrombin time (PT) or International Normalised Ratio (INR) ≤1.5 x ULN

Exclusion Criteria:

1. Nodule adjacent to or encircling a large mediastinal vessel (e.g., aorta, superior vena cava, main pulmonary artery, main pulmonary vein, etc.), with a distance from the vessel <5 mm;
2. Subpleural nodules (<5 mm from the pleura);
3. patients with regional lymph node metastasis or distant metastasis confirmed by chest enhanced CT/HRCT;
4. patients with severe bleeding tendency, coagulation dysfunction that cannot be corrected within a short period of time (prothrombin time >18 s, prothrombin activity <40%) and/or platelet count <50 × 109/L;
5. severe interstitial pneumonia, severe pulmonary fibrosis or severe emphysema;
6. malignant pleural effusion;
7. treatment for the following:

   * received systemic anti-tumour therapy such as chemotherapy, targeted therapy, immunotherapy, etc;
   * Received any investigational drug therapy;
   * High dose immunosuppressive drugs (systemic glucocorticoids greater than 10mg/day prednisone or its equivalent) within 4 weeks prior to the entry assessment;
   * Received a live attenuated vaccine within 4 weeks prior to the entry assessment (or plan to receive a live attenuated vaccine during the study period);
   * Major surgery (e.g., open heart, open chest, or open abdomen) or unhealed surgical wounds, ulcers, or fractures within 4 weeks prior to the enrolment assessment;
8. Have another uncontrolled serious medical condition, including but not limited to:

   * Serious infections that are active or not well controlled clinically;
   * HIV infected (HIV antibody positive);
   * Acute or chronic active hepatitis B (HBV DNA positive) or acute or chronic active hepatitis C (HCV antibody positive);
   * Active tuberculosis, etc;
   * Class III-IV congestive heart failure (New York Heart Association classification) with poorly controlled and clinically significant arrhythmias;
   * Uncontrolled arterial hypertension (systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg);
   * Any arterial thrombosis, embolism or ischaemia such as myocardial infarction, unstable angina pectoris, cerebrovascular accident or transient ischaemic attack within 6 months prior to enrolment for treatment;
   * Diseases requiring anticoagulant therapy with Favalin (Coumadin);
   * Uncontrolled hypercalcaemia (greater than 1.5 mmol/L Ca2+ or calcium greater than 12 mg/dL or corrected serum calcium greater than ULN) or symptomatic hypercalcaemia requiring continued bisphosphonate therapy;
   * concomitant other malignancies (except those that have been eradicated, e.g., carcinoma in situ of the uterine cervix, non-melanoma skin cancer, etc.); and
9. Other acute or chronic medical conditions, psychiatric disorders, or abnormal laboratory test values that may result in: increased risk associated with study participation or administration of study medication, or interference with the interpretation of study results, and that, in the investigator's judgement, classifies the patient as ineligible for participation in this study;
10. Pregnant or lactating females.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with high-risk lung nodules/early stage lung cancer
Sampling Method: Probability Sample
Enrollment: 656 (Estimated)
Dates: Start 2025-04-12 (Actual); Primary Completion 2028-12-21 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
relapse-free survival, RFS | Three years, five years
  Time from grouping to relapse or death from any cause or last contact with a surviving patient (whichever occurs first).

SECONDARY OUTCOMES:
Technical success rate | Perioperative/Periprocedural
  1. When the tumour is treated according to a predetermined protocol with complete overlap of the ablation area (ablation border > tumour border by at least 5 mm), the operation is defined as a technical success when imaging follow-up demonstrates complete macroscopic ablation of the tumour, and technical success is defined as the percentage of the calculation of technical success.
Pulmonary Function Assessment | Baseline, 1 month, 3 months, 6 months, 12 months.
  The process of quantitatively analysing and comprehensively evaluating the functional status of the patient's lungs, such as ventilation and gas exchange, by measuring the patient's first-second force expiratory volume (FEV1) and forceful lung capacity (FVC).
overall survival, OS | Three years, five years
  Time from grouping to death from any cause or last contact with surviving patient (whichever occurs first).
local regional resection, LRR | Within five years
  Proportion of tumours with cancer metastases reappearing at the primary site or elsewhere within the same lobe of the lung or in the lung or draining hilar lymph nodes after receiving treatment.
Security Indicators | Within six months after surgery
  Adverse event rates, and operation-related adverse event rates throughout the study: adverse events occurring within 30 days of ablation treatment and operation-related adverse events of surgical treatment (AE&SAE), evaluated according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0.

OTHER OUTCOMES:
Biological indicators of peripheral blood | Baseline AND 1 month
  Methylation results of lung cancer-related genes
Quality of life score | Baseline AND 6 months
  Scored on a questionnaire, the higher the score the better the quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Chengzhi Zhou, Doctor, Study Director — Guangzhou Institute of Respiratory Disease (Responsible Party)
Locations (1):
- Guangzhou Institute of Respiratory Disease (Responsible Party), Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided